CLINICAL TRIAL: NCT01444157
Title: Family and Coping Oriented Palliative Homecare Nursing as a Supplement to Standard Homecare Nursing Aimed at Advanced Cancer Patients - a Randomized Intervention Trial
Brief Title: Family and Coping Oriented Palliative Homecare Nursing Aimed at Advanced Cancer Patients
Acronym: FamCope
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Collaborators: Danish Cancer Society (Other); Lundbeck Foundation (Other); Sygekassernes Helsefond (Other); The Novo Nordic Foundation (Other); Danish Nurses Organisation (Other); Danish Regions (Unknown)
Responsible Party: Principal Investigator, Anne Birgitte Hjuler Ammari, Principal investigator, Bispebjerg Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: FamCope2011
Record Dates: First submitted 2011-09-29; First posted 2011-09-30 (Estimated); Last update posted 2014-07-18 (Estimated); Status verified 2014-07

CONDITIONS: Advanced Cancer
MeSH Terms: interventions — Palliative Care; Coping Skills; Quality of Life; Needs Assessment; Patient Readmission

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Palliative homecare nursing group (Experimental): In addition to the standard homecare nursing the families will receive six home visits from a research nurse with at least 1 year specialised palliative care experience. During the first 2 hour visit a family assessment is obtained containing identification of family roles, resources and coping strategies. The first home visit takes place no later than one week after randomization. The visits continues every third week up to 16 weeks, each visit with a duration of 1,5 hours. At every visit the EORTC-QLQ-C30 patient administered questionnaire is used to identify the nature, frequency and intensity of the patients physical and psychosocial problems.
  Interventions: Other: Palliative homecare nursing
- Standard homecare nursing group (No Intervention): Patients continue to receive the standard homecare nursing. They can contact municipality services for visitation to homecare nursing if they feel that additional homecare is needed or if they do not yet receive this service and feel they need homecare nursing.

INTERVENTIONS:
Other: Palliative homecare nursing — The nurse helps the family assess the identified problems. Written coping strategies according to each problem is produced including actions of the patient, family member, nurse or others. At the same time the nurse keeps attention to the family members specific needs of knowledge and support when handling direct or indirect care, understanding and coping with the disease, treatment, physical, psychosocial and economical problems and the family members own physical and mental health. The nurse provides knowledge to the family on how to prevent and/or cope with problems that may occur or re-occur and/or accepts or adapt to unsolvable problems.
  Other Names: Palliative care; Advanced cancer; Family nursing; Community nursing; Coping; Quality of life; Needs assessment; Family satisfaction; Hospital readmission
  Arms: Palliative homecare nursing group

SUMMARY:
When facing life threatening illness such as advanced cancer palliative care is needed to improve quality of life of patients and their families through the prevention and relief of suffering. Palliative care at an early stage prevents the development of problems and symptoms, but time, resources and experience are needed in the primary care sector in Denmark to deal with the problems families experiencing life with advanced cancer are facing. The aims of this study are to test, evaluate and further develop interventions that can help identify and assess problems, resources and opportunities of families experiencing life with advanced cancer, and on this background to help the families cope with their situation in cooperation with healthcare professionals to an extent where the family's quality of life increases, their physical and psychosocial problems are relieved, their symptoms of anxiety and depression are reduced, family satisfaction with health professionals are increased and acute readmissions to hospital are prevented.

DETAILED DESCRIPTION:
Screening for patients will take place in the oncological, gynecological medical, surgical departments of three hospitals in Copenhagen, Denmark among patients diagnosed with cancer. Patients eligible for the study will be informed about the study during hospital admission and asked to participate together with a close relative/family member. When written informed consent has been obtained from both patient and relative they will be asked to fill in questionnaires with background information about sociodemographic data, their physical and psychosocial functioning and quality of life EORTC (QLQ-C30/patient and SF36/relative), their symptoms of anxiety and depression (HAD Scale/patient and relative) and family satisfaction with health care professionals(FamCare/relative). When patients have been discharge from hospital to their own home the families are randomized to control or intervention group. First visit from the research nurse takes place no later than one week after randomization. Visits takes place week 1,4,7,10,13 and 16 after randomization. The questionnaires EORTC QLQ-C30 (patient), HAD Scale (patient and relative), SF 36 (relative) and FamCare (relative) are mailed by post to the families to be answered at week 9, 16 and 24 after randomization. Information about the amount of care the family receives from the municipality (standard homecare) will be obtained from municipal registers. Information about readmissions to hospital are obtained from hospital registers.

The research nurses has a minimum of one year experience within specialised palliative care. The nurses has also participated in a two day course on how to produce and utilise family assessment and have been introduced to the background theory on coping and family nursing.

ELIGIBILITY:
Inclusion Criteria:

At least one of the following

* Cancer stage 3 or 4 (according to hospital journal)and at least one treatment after relapse without satisfying effect on the disease
* The patient is aware that further treatment is of palliative or life prolonging nature

And also all of following inclusion criterions

* The patient has a family member that would like to participate (The family member must be involved in the patients care at least two times a week)
* At least 18 years old (patient and family member)
* Understand and speak danish (patient and family member)
* Live in the area of the municipalities of Copenhagen or Frederiksberg
* Discharge from hospital to own home
* Written informed consent (patient and family member)

Exclusion Criteria:

* Terminal fase of disease
* Contact with specialised palliative care
* Incapable of co-operating with trial protocol
* Participant in another behavioral intervention study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2011-10; Primary Completion 2013-10 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Patient reported health related quality of life | Baseline, week 9, week 16 and week 24
  The change in mean scores from baseline to each follow up as measured in the Quality of life questionnaire EORTC QLQ-C30 scale score(Developed by the European Organization for Research and Treatment of Cancer)in relation to the Global health status scale.

SECONDARY OUTCOMES:
Patient reported symptoms and problems | Baseline, week 9, week 16 and week 24
  The change in mean scores from baseline to each follow up as measured in the EORTC QLQ-C30 questionnaire scale score in relation to its functional scales and symptom scales/items.
Patients symptoms of anxiety and depression | Baseline, week 9, week 16 and week 24
  The change in mean scores from baseline to each follow up according to the HADS questionnaire (Hospital Anxiety and Depression Scale) Scores are self-reported.
Family members symptoms of anxiety and depression | Baseline, week 9, week 16, week 24 and 12 months
  The change in mean scores from baseline to each follow up according to the HADS questionnaire. Scores are self-reported.
Family members health related quality of life | Baseline, week 9, week 16, week 24 and 12 months
  The change in mean scores from baseline to each follow up. Scores are self-reported and measured in the SF36 v1 questionnaire.
Family satisfaction with the health care services provided to the patient | Baseline, week 9, week 16, week 24 and 12 months
  The change in mean scores from baseline to each follow up. Scores are self-reported and measured in the FAMCARE questionnaire
Acute readmission to hospital | week 16 and 24
  The change in mean number of acute readmissions and mean period of hospitalizations (measured in days) from inclusion to the study to week 16 and 24. Readmissions must be related to the patients cancer disease

CONTACTS AND LOCATIONS:
Overall Officials: Susan Rydahl Hansen, Cand.cur, PhD, Study Director — Research Unit of Clinical Nursing, Bispebjerg Hospital; Anne Birgitte Hjuler Ammari, Cand.scient.san, Principal Investigator — Research Unit of Clinical Nursing, Bispebjeg Hospital
Locations (3):
- Denmark (3):
  - Frederiksberg Hopsital, Copenhagen, Frederiksberg
  - Bispebjerg Hospital, Copenhagen, NV
  - Rigshospitalet, Copenhagen